CLINICAL TRIAL: NCT01913314
Title: Disposition of [^14C]-LY2835219 Following Oral Administration in Healthy Subjects
Brief Title: A Study of Carbon-14-Labeled LY2835219 ([^14C]-LY2835219) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14930; I3Y-MC-JPBD (Other: Eli Lilly and Company)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [^14C]-LY2835219 (Experimental): Single 150 milligram (mg) oral dose solution of LY2835219 containing 5 micro-curies of (µCi) [^14C] labeled drug
  Interventions: Drug: [^14C]-LY2835219

INTERVENTIONS:
Drug: [^14C]-LY2835219 — Administered as oral solution
  Other Names: abemaciclib

SUMMARY:
This type of study is called a radiolabeled study. For this study, LY2835219 (study drug) has been specially prepared to contain radiolabeled carbon [^14C]. [^14C] is a naturally occurring radioactive form of the element carbon. This study will help understand how the drug appears in the blood, urine, and stool after it is administered.

In addition, this study will also evaluate the safety and tolerability of a single dose of LY2835219 when given to healthy participants. Information about any side effects that may occur will also be collected.

This study will last about 3 weeks for each participant, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male or female participants as determined by medical history and physical examination
* Male participants will be sterile
* Female participants will be surgically sterile or postmenopausal
* Have a body mass index (BMI) of 18 to 29 kilograms per square meter (kg/m^2)
* Have venous access sufficient to allow for blood sampling

Exclusion Criteria:

* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Gastrointestinal disorders causing clinically significant symptoms such as nausea, vomiting, and diarrhea, or malabsorption syndromes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- [^14C]-LY2835219: Single 150-milligram (mg) LY2835219 dose containing 5 micro- curies (µCi) of carbon-14-labeled LY2835219 ([^14C]-LY2835219), administered as an oral solution.
Period: Overall Study
Arm/Group | [^14C]-LY2835219
Started | 6
Received Study Drug | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who received study drug.
Groups:
- [^14C]-LY2835219: Single 150-mg LY2835219 dose containing 5 µCi of [^14C]-LY2835219, administered as an oral solution.
Arm/Group | [^14C]-LY2835219
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Urinary and Fecal Excretion of LY2835219-Related Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Description: The percentage of the total radioactive dose administered that was excreted in urine or feces = (amount of radioactive dose recovered in urine or feces / total radioactive dose administered) * 100.
Time Frame: Predose up to Day 14 postdose; Fecal samples collected at 24-hour (h) intervals; Urine collected at 0 to 6 h, 6 to 12 h, and 12 to 24 h postdose and at 24-h intervals thereafter up to Day 14 postdose
Population: Participants who received study drug.
Measure: Mean (Standard Deviation); unit: percentage radioactive dose administered
Arm/Group | [^14C]-LY2835219
Number analyzed (Participants) | 6
percentage radioactive dose administered
  Urine | 3.43 (2.20)
  Feces | 81.0 (6.71)

2. Secondary Outcome: Plasma Pharmacokinetics (PK) of LY2835219 and Metabolite of LY2835219: Maximum Observed Concentration (Cmax)
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 h postdose, thereafter at 24-h intervals up to Day 14 postdose
Population: Participants who received study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | [^14C]-LY2835219
Number analyzed (Participants) | 6
nanograms per milliliter (ng/mL)
  LY2835219 | 63.7 (49)
  M20 | 30.9 (19)

3. Secondary Outcome: Plasma PK of Radioactivity: Cmax
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 h postdose, thereafter at 24-h intervals up to Day 14 postdose
Population: Participants who received study drug and had evaluable PK Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalents per gram (ng Eq/g)
Arm/Group | [^14C]-LY2835219
Number analyzed (Participants) | 6
nanogram equivalents per gram (ng Eq/g) | 123 (27)

4. Secondary Outcome: Plasma PK of LY2835219, Metabolite of LY2835219, and Radioactivity: Time of Maximum Observed Concentration (Tmax)
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 h postdose, thereafter at 24-h intervals up to Day 14 postdose
Population: Participants who received study drug and evaluable PK tmax data.
Measure: Median (Full Range); unit: h
Arm/Group | [^14C]-LY2835219
Number analyzed (Participants) | 6
h
  LY2835219 | 8.00 [6.00 to 8.00]
  M20 | 8.00 [6.00 to 10.00]
  Total Radioactivity | 8.00 [6.00 to 10.00]

5. Secondary Outcome: Plasma PK of LY2835219 and Metabolite of LY2835219: Area Under the Concentration-Time Curve From Time Zero to the Last Time Point With a Measurable Concentration [AUC(0-tlast)]
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 h postdose, thereafter at 24-h intervals up to Day 14 postdose
Population: Participants who received study drug and had evaluable PK AUC(0-tlast) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | [^14C]-LY2835219
Number analyzed (Participants) | 6
nanograms*hour/milliliter (ng*h/mL)
  LY2835219 | 2310 (85)
  M20 | 1760 (43)

6. Secondary Outcome: Plasma PK of Radioactivity: AUC(0 to Tlast)
Description: The PK of radioactivity was measured as nanogram equivalents times hours per gram (ng Eq*h/g).
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 h postdose, thereafter at 24-h intervals up to Day 14 postdose
Population: Participants who received study drug and had evaluable PK AUC(0-tlast) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng Eq*h/g
Arm/Group | [^14C]-LY2835219
Number analyzed (Participants) | 6
ng Eq*h/g | 6580 (41)

7. Secondary Outcome: Plasma PK of LY2835219 and Metabolite of LY2835219: Area Under the Concentration Versus Time Curve From Zero to Infinity [AUC(0-∞)]
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 h postdose, thereafter at 24-h intervals up to Day 14 postdose
Population: Participants who received study drug and had evaluable PK AUC(0-∞) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | [^14C]-LY2835219
Number analyzed (Participants) | 6
ng*h/mL
  LY2835219 | 2370 (83)
  M20 | 1830 (42)

8. Secondary Outcome: Plasma PK of Radioactivity: AUC(0-∞)
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 h postdose, thereafter at 24-h intervals up to Day 14 postdose
Population: Participants who received study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng Eq*h/g
Arm/Group | [^14C]-LY2835219
Number analyzed (Participants) | 6
ng Eq*h/g | 7010 (42)

9. Secondary Outcome: Relative Abundance of LY2835219 and Metabolites of LY2835219 Eliminated in Urine and Feces
Description: The abundance (as percentage dose) of LY2835219 or its metabolites eliminated in feces is calculated as = (amount of LY2835219 or its metabolites recovered in feces / total amount administered) * 100. Due to low radioactivity of dose recovered in urine, further quantitative profiling of urine was not conducted.
Time Frame: Predose through 216 h postdose; Fecal samples collected at 24-h intervals
Population: Participants who received study drug and had evaluable PK data. No participants were analyzed for relative abundance of LY2835219 and metabolites of LY2835219 in urine.
Measure: Number; unit: percentage of radioactive dose excreted
Arm/Group | [^14C]-LY2835219
Number analyzed (Participants) | 6
percentage of radioactive dose excreted
  LY2835219 | 7
  Metabolites | 52

10. Secondary Outcome: Relative Abundance of LY2835219 and Metabolites of LY2835219 in Plasma
Description: The relative abundance of LY2835219 or its metabolites in plasma were estimated based on AUC(0-∞) and reported as a percentage of total plasma radioactivity. The relative abundance of LY2835219 or its metabolites calculated as = [AUC (0-∞) of LY2835219 or its metabolites in plasma / AUC (0-∞) of total plasma radioactivity] * 100.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 h postdose, thereafter at 24-h intervals up to Day 14 postdose
Population: Participants who received study drug and had evaluable PK AUC(0-∞) data.
Measure: Number; unit: percentage of total plasma radioactivity
Arm/Group | [^14C]-LY2835219
Number analyzed (Participants) | 6
percentage of total plasma radioactivity
  LY2835219 | 34
  Metabolites | 44

ADVERSE EVENTS:
Arm/Group | [^14C]-LY2835219
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [^14C]-LY2835219 (N=6)
Vessel Puncture Site Haematoma (General disorders) | 2 (2)
Vessel Puncture Site Pain (General disorders) | 1 (1)
Vessel Puncture Site Swelling (General disorders) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days